CLINICAL TRIAL: NCT03967379
Title: Multimodal Mobile Intervention Application (App) to Address Sexual Dysfunction in Hematopoietic Stem Cell Transplant Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-104
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Other Cancer
Keywords: Other Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile app plus enhanced standard care (Experimental): * Patients will received enhanced standard care in addition to access to the sexual health mobile app.
  * The app will also prompt patients to engage their partners with specific exercises.
  Interventions: Behavioral: Mobile App + enhanced standard care; Other: Enhanced Standard Care
- Enhanced Standard Care (Other): * Patients will receive Enhanced Standard Care
  * Patients will meet with a transplant clinician for a brief medical examination to assess the need for medications for erectile dysfunction, vaginal atrophy, or vulvovaginal GVHD
  * Patients will not have access to the sexual health mobile app
  Interventions: Other: Enhanced Standard Care

INTERVENTIONS:
Behavioral: Mobile App + enhanced standard care — An intervention to help address sexual dysfunction among HCT survivors
  Arms: Mobile app plus enhanced standard care
Other: Enhanced Standard Care — Standard of care administered by the institution

SUMMARY:
This research study is being done to evaluate whether the use of a mobile app can help transplant survivors experiencing sexual health problems.

DETAILED DESCRIPTION:
Frequently survivors of stem cell transplantation report significant problems with their sexual function that impacts their quality of life, mood, and their intimacy and relationship with their partners. These issues can be very distressing to patients and their loved ones. The study doctors want to know if the use of a mobile app intervention focused on improving sexual function may improve participants overall care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) who underwent an autologous or allogeneic HCT at least 3 months prior to study enrollment.
* Ability to speak English or able to complete questionnaires with assistance required from an interpreter or family member.
* Positive screen for sexual dysfunction that is causing distress based on the NCCN survivorship guidelines

Exclusion Criteria:

* Recurrent disease requiring treatment
* Significant uncontrolled psychiatric disorder (psychotic disorder, bipolar disorder, major depression) or other co-morbid disease (dementia, cognitive impairment), which the treating clinician believes prohibits the ability to participate in study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Groups:
- Mobile App Plus Enhanced Standard Care: * Patients will received enhanced standard care in addition to access to the sexual health mobile app.
  * The app will also prompt patients to engage their partners with specific exercises.
  Mobile App + enhanced standard care: An intervention to help address sexual dysfunction among HCT survivors
  Enhanced Standard Care: Standard of care administered by the institution
- Enhanced Standard Care: * Patients will receive Enhanced Standard Care
  * Patients will meet with a transplant clinician for a brief medical examination to assess the need for medications for erectile dysfunction, vaginal atrophy, or vulvovaginal GVHD
  * Patients will not have access to the sexual health mobile app
  Enhanced Standard Care: Standard of care administered by the institution
Period: Overall Study
Arm/Group | Mobile App Plus Enhanced Standard Care | Enhanced Standard Care
Started | 30 | 30
Completed | 24 | 22
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile App Plus Enhanced Standard Care | Enhanced Standard Care | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Full Range); unit: Years] | 54.5 [24.3 to 75] | 57.7 [27.9 to 77] | 57.2 [24.3 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 18 | 18 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 29 | 57
  Black | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Based on Proportion of Subjects Enrolled
Description: feasibility will be a priori defined as at least 60% o eligible patients enrolled in the study.
Time Frame: 2 years
Population: This is the total number of patients identified as eligible for the study (to reflect feasibility metric)
Measure: Count of Participants; unit: Participants
Groups:
- Total Study Sample: The entire cohort
Arm/Group | Total Study Sample
Number analyzed (Participants) | 95
Participants | 60

2. Secondary Outcome: Compare Patient-reported Global Satisfaction With Sex (PROMIS Sexual Function and Satisfaction Measure) Between the Study Groups
Description: patient-reported global satisfaction using the PROMIS Sexual Function and Satisfaction Measure. Higher scores indicate better global satisfaction with sex (raw score range 4-25). We will use raw score for reporting in this study given the extent of illness in this population.
Time Frame: 8 weeks
Population: comparison of outcomes at week-8
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mobile App Plus Enhanced Standard Care | Enhanced Standard Care
Number analyzed (Participants) | 30 | 30
score on a scale | 14.6 [12.8 to 16.4] | 12.3 [10.5 to 14.1]

3. Secondary Outcome: Compare Patient-reported Interest in Sexual Activity (PROMIS Sexual Function and Satisfaction Measure - Interest in Sexual Activity Domain) Between the Study Groups
Description: compare patient-reported interest in sexual activity using the PROMIS Sexual Function and Satisfaction Measure - Interest in Sexual Activity Domain). higher score indicate better interest in sex (raw score range 2-10).
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mobile App Plus Enhanced Standard Care | Enhanced Standard Care
Number analyzed (Participants) | 30 | 30
score on a scale | 6.70 [6.1 to 7.4] | 5.7 [5 to 6.4]

4. Secondary Outcome: Compare Patient-reported Orgasm (PROMIS Sexual Function and Satisfaction Measure - Orgasm Domain) Between the Study Groups
Description: compare patient-reported orgasm using the PROMIS Sexual Function and Satisfaction Measure - Orgasm Domain). higher score indicate better orgasm (raw score range 3-15).
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mobile App Plus Enhanced Standard Care | Enhanced Standard Care
Number analyzed (Participants) | 30 | 30
score on a scale | 9.7 [8.4 to 10.8] | 8.3 [7.0 to 9.5]

5. Secondary Outcome: For Males: Compare Patient-reported Erectile Function (PROMIS Sexual Function and Satisfaction Measure - Erectile Function Domain) Between the Study Groups
Description: for males: compare patient-reported erectile function using the PROMIS Sexual Function and Satisfaction Measure - Erectile Function Domain). higher score indicate better erectile function (raw score range 0-55)
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mobile App Plus Enhanced Standard Care | Enhanced Standard Care
Number analyzed (Participants) | 18 | 18
score on a scale | 36.6 [30.2 to 42.9] | 27.9 [21.3 to 34.5]

6. Secondary Outcome: For Females: Compare Patient-reported Lubrication and Vaginal Comfort (PROMIS Sexual Function and Satisfaction Measure - Lubrication and Vaginal Comfort Domains) Between the Study Groups
Description: For females: compare patient-reported vaginal comfort and lubrication using the PROMIS Sexual Function and Satisfaction Measure- Lubrication and Vaginal Comfort Domain). higher score indicate better lubrication (raw score 0-25)
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mobile App Plus Enhanced Standard Care | Enhanced Standard Care
Number analyzed (Participants) | 12 | 12
score on a scale | 13.5 [10.4 to 16.4] | 12.1 [9.3 to 14.9]

7. Secondary Outcome: Compare Patient Reported Quality of Life (FACT-BMT) Between the Study Groups
Description: compare patient-reported quality of life using the Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT). higher score indicate better quality of life (range 0-196)
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mobile App Plus Enhanced Standard Care | Enhanced Standard Care
Number analyzed (Participants) | 30 | 30
score on a scale | 115.6 [110.8 to 120.4] | 108.3 [103.3 to 113.2]

8. Secondary Outcome: Compare Patient Reported Depression Symptoms (HADS-depression) Between the Two Study Groups
Description: compare patient-reported depression symptoms using Hospital Anxiety and Depression Scale (HADS-Depression). higher subscale score indicate worse depression symptoms (range 0-21)
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mobile App Plus Enhanced Standard Care | Enhanced Standard Care
Number analyzed (Participants) | 30 | 30
score on a scale | 3.6 [2.6 to 4.6] | 5.4 [4.3 to 6.4]

9. Secondary Outcome: Compare Patient Reported Anxiety Symptoms (HADS-anxiety) Between the Two Study Groups
Description: compare patient-reported depression symptoms using Hospital Anxiety and Depression Scale (HADS-Anxiety). higher subscale score indicate worse anxiety symptoms (range 0-21)
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mobile App Plus Enhanced Standard Care | Enhanced Standard Care
Number analyzed (Participants) | 30 | 30
score on a scale | 4.5 [3.3 to 5.7] | 6.4 [5.1 to 7.7]

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored and assessed as part of this protocol given that this is a supportive care trial in a population at high risk for death and illness due to their underlying disease,
Description: Adverse events were not monitored and assessed as part of this protocol given that this is a supportive care trial in a population at high risk for death and illness due to their underlying disease,
Arm/Group | Mobile App Plus Enhanced Standard Care | Enhanced Standard Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT03967379/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT03967379/ICF_001.pdf